CLINICAL TRIAL: NCT00475189
Title: Prospective Comparison of Hormone Withdrawal Symptoms of a 24/4 Regimen With a 21/7 Regimen of OC
Brief Title: Study of Loestrin 24(24 Days of "Real" Pills) Fe Versus Loestrin 1/20 (21 "Real" Pills)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Warner Chilcott (Industry)
Responsible Party: Dr. Patricia Sulak, Scott and White Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 60783
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Pelvic Pain; Headaches; Emotional
Keywords: birth control; PMS; headaches; mood swings; pelvic pain
MeSH Terms: conditions — Pelvic Pain; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: loestrin 24/4 vs loestrin 1/20
- II (Active Comparator): loestrin 1/20 given 1 tab 21/7
  Interventions: Drug: loestrin 1/20

INTERVENTIONS:
Drug: loestrin 24/4 vs loestrin 1/20 — One month of loestrin 1/20 then randomized to Loestrin 24/4 or Loestrin 1/20 x 3 months. After 3 months if randomized to 1/20 will be switched to 24/4 if already on 24/4 will be given a choice which OC they want to continue for 3 more months.
  Other Names: Brand name for Loestrin FE 1/20 is Junel FE and Microgestin FE.
  Arms: 1
Drug: loestrin 1/20 — loestrin 1/20 1 tab 21/7 x 3mo and then changed to Loestrin 24 FE
  Other Names: Junel FE; Microgestin FE
  Arms: II

SUMMARY:
The purpose of this research study is to assess hormone withdrawal symptoms in women while taking an oral contraceptive in the novel 24/4 (24 days of "real" pills) manner in comparison to taking pills in the standard 21/7 (21 "real" pills) manner.

It is hypothesized that the 24/4 method will reduce common hormone withdrawal symptoms compared to the standard 21/7 regimen.

It is further hypothesized that women using the 24/4 regimen will report greater satisfaction scores.

DETAILED DESCRIPTION:
Women who will be considered for this study are those who are presently taking combination estrogen/progestin contraception for at least 2 months. They must be between the ages of 18 and 48 years with a body mass index of 40 or less. Study participants will be asked to keep a daily diary of symptoms based on the symptoms listed above. This requires ranking the severity of bleeding, pelvic pain, mood, and headaches based on a scale defined on the daily diary. All subjects will keep track of any pain medication that they take on a medication log.

Subjects that are not sure if their symptoms (mood, pelvic pain or headache) increase on days 1-3 and 18-28, will be asked to keep the diary while taking their current contraceptive medication. After they record their symptoms in the diary, it will be evaluated by the study coordinator to see if they qualify (which means that mood, pelvic pain and headache must have increased on days 1-3 and 18-28 compared to days 4-17). If they qualify, visit 1 will be scheduled.

At visit 1, subjects will undergo a physical exam and a pelvic exam. Subjects may be required to have a Pap smear if one has not been performed or if there is not sufficient documentation of one within the past year. Subjects will be given a single pack of Loestrin 1/20 for cycle #1 along with their symptoms calendars and medication log.

All women will begin the study with one month of Loestrin 1/20, to be taken in a normal 21/7 manner, and will complete a daily questionnaire. To continue in the study, subjects must be classified as having substantial fluctuation in their symptoms. At visit 2, (end of cycle #1), subjects will return their completed calendar to the study coordinator. The calendar will be reviewed for compliance and for eligibility based on symptom criteria. Subjects will also be scheduled for lab work. Women who continue in the study will be randomly assigned either to a group to start taking Loestrin 24 Fe (24 real pills and 4 placebo pills - Group 1), or to a group to continue taking Loestrin 1/20 in the standard 21/7 fashion for an additional 3 cycles (Group 2). All women will be asked to continue keeping a daily log of their symptoms, which will be turned in to the study coordinator at each of the scheduled visits.

Subjects will not be given the choice initially as to which group they will be placed; however all women will be given the opportunity to evaluate the 24/4 regimen. After the first 3 randomized cycles (visit 3), subjects will turn in their calendars to the study coordinator. Group 1 will be given a choice between continuing Loestrin 24 Fe or going back to Loestrin 1/20. Group 1 will complete a brief survey regarding their choice and will be given 3 packs of the pill of choice. All Group 2 subjects will be switched onto 3 cycles of Loestrin 24 Fe. Subjects in both groups will continue keeping their daily symptoms calendar.

At visit 4, the end of cycle #5, all subjects will turn in their calendars to the study coordinator.

At visit 5, the end of cycle #7, subjects will turn in their calendars to the study coordinator. All subjects will fill out a questionnaire. Subjects will be evaluated and will be given a prescription for the OC of their choice.

Subjects will also be asked to complete mid-study and end of study quality of life and satisfaction questionnaires.

Blood Draws 1-8 One of the objectives of this study is to compare hormone withdrawal symptoms with actual hormone levels. Measuring hormones requires samples of blood. Over the course of the study, there will be a total of 8 separate blood samples (for a total of approximately 8 teaspoons of blood) to be taken from each subject. Subjects in Group 1 who were randomized to Loestrin 24 Fe during cycles 2 through 4 will start blood sampling on cycle day 24, the last day of active pills in this cycle and continue at three day intervals. Subjects in Group 2 who were randomized to Loestrin 1/20 during cycles 2 through 4 will start blood sampling on cycle day 21, the last day of active pills in the 4th cycle and continue at three day intervals.

ELIGIBILITY:
Inclusion Criteria:

* current users (>2 months) of a combination hormonal contraceptive (OC, contraceptive ring, contraceptive patch) with at least the most recent cycle ending with a 7 day HFI
* age 18-48
* BMI of 40 or less
* not desiring to become pregnant during the study time (about 8 months)
* capable and reliable in regards to recording and maintaining a daily symptoms log

Exclusion Criteria:

* a condition which will not allow you to use combination hormonal contraception; including a past or present history of diabetes, high blood pressure, stroke, breast cancer, heart attacks, blood clots, liver disease, or systemic lupus erythematosus.
* are pregnant or plan to become pregnant in the next 8 months or while you are in the study.
* a smoker greater than or equal to 35 years of age. You smoke 10 or more cigarettes a day and you are under the age of 35.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Use of the Scott and White (S&W) Daily Symptoms Calendar, which records patient's subjective rating of mood, pelvic pain, flow, headache, and number and dose of pain medicines taken. | 8 months
Measuring the levels of endogenous hormone (estradiol) in order to correlate serum estradiol levels with withdrawal symptoms during and after the two OC types (4-days versus 7-days) of hormone free intervals. | one month

SECONDARY OUTCOMES:
satisfaction Surveys | given midway through the study and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sulak, MD, Principal Investigator — Scott and White Hospital & Clinic
Locations (1):
- Scott & White Hospital and Clinic, Temple, Texas, United States